CLINICAL TRIAL: NCT07093606
Title: Eltrombopag Induced Liver Dysfunction During Treatment of Immunethrombocytopenic Purpura
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Peter Adel Alfy, Resident , Internal medicine, Faculty of Medicine Sohag university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Soh-Med--25-7-4MS
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: ITP - Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- this group will receive Eltrombopag tabelts (Experimental): ITP patients in this group receive Eltrombopag then follow up by liver functions test to evulate occurance of liver disorders .
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — ITP patients will receive Eltrombopag and evulate occurance of liver disordres .

SUMMARY:
this study amis to assess the incidence and severity of liver dysfunction in ITP patients receiving eltrombopag.

ELIGIBILITY:
Inclusion Criteria Adult patients (≥18 years) diagnosed with primary ITP. Receiving eltrombopag as part of their treatment. Baseline liver function tests (LFTs) within normal limits. Patients with diabetes Patients without diabetes Patients with fatty liver Patients without fatty liver

Exclusion Criteria:

Pre-existing liver disease (e.g., hepatitis, cirrhosis, NAFLD). Concurrent use of hepatotoxic drugs. Patients lost to follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
•To assess the incidence and severity of liver dysfunction in ITP patients receiving eltrombopag. | 3-6 months after receiving eltombopag
  the incidence and severity of liver dysfunction in ITP patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

REFERENCES:
- [Background] Bidika E, Fayyaz H, Salib M, Memon AN, Gowda AS, Rallabhandi B, Cancarevic I. Romiplostim and Eltrombopag in Immune Thrombocytopenia as a Second-Line Treatment. Cureus. 2020 Aug 21;12(8):e9920. doi: 10.7759/cureus.9920. PMID 32968581
- [Background] Kuter DJ. New thrombopoietic growth factors. Blood. 2007 Jun 1;109(11):4607-16. doi: 10.1182/blood-2006-10-019315. Epub 2007 Feb 8. PMID 17289815
- [Background] Ptushkin VV, Vinogradova OY, Pankrashkina MM, Chernikov MV, Arshanskaya EG, Tkachenko NE. Thrombopoietin Receptor Agonists in the Treatment of Chronic Resistant Primary Immune Thrombocytopenia: Efficacy and Safety Data in Real Clinical Practice. Ter Arkh. 2018 Aug 17;90(7):70-76. doi: 10.26442/terarkh201890770-76. PMID 30701925